CLINICAL TRIAL: NCT03166670
Title: Parasitic Causes of Secretory Diarrhea in Children and Chronically Ill Adult.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Elderwy, Principal Investigator, Assiut University
Other Study IDs: PSDCC
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Diarrhea, Secretory
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: children with acute secretory diarrhea
  Interventions: Diagnostic Test: stool examination; Diagnostic Test: real time polymerase chain reaction
- Control group: normal healthy children
  Interventions: Diagnostic Test: stool examination; Diagnostic Test: real time polymerase chain reaction

INTERVENTIONS:
Diagnostic Test: stool examination — collection of stool specimen and microscopic examination for parasites
Diagnostic Test: real time polymerase chain reaction — evaluation of genotype of cryptosporidium in stool specimen

SUMMARY:
Diarrhea is one of the most common reasons for people to seek medical advice - but it can range from being a mild, temporary condition, to be life threading condition. It is estimated that there are 2 billion cases of diarrheal disease every year globally, and that 1.9 million children below the age of 5 years, mostly in developing countries, die annually.

DETAILED DESCRIPTION:
Secretory diarrhea has many causes as infection with bacteria, viruses or protozoa. It results from increased chloride secretion, decreased sodium absorption, or increased mucosal permeability . Parasitic pathogens induce Secretory diarrhea as they infect and damage the absorptive villus tips, leaving Secretory crypts unbalanced, to cause net secretion and diarrhea. Parasitic causes include Cryptosporidium parvum or hominis ,Capillaria philippinensis and Giardia lamblia. Cryptosporidiosis is also recognized as a cause of prolonged and persistent diarrhea in children and persons with impaired immunity. The disease is transmitted via the fecal-oral route from infected hosts. It can be also transmitted following animal contact, ingestion of water (mainly during swimming), or through food. Cryptosporidium has emerged as the most frequently recognized cause of water-associated outbreaks of gastroenteritis. This is because of the oocyst stage in its life cycle; Cryptosporidium can resist disinfection, including chlorination, and can survive for a prolonged period in the environment.

ELIGIBILITY:
Inclusion Criteria:

1. Children presented with secretory diarrhea(acute watery diarrhea) attend to out clinic lab of Assiut University pediatric hospital or admitted in pediatric hospital(gastroenterology department) during the study period.
2. adult patients having acute watery diarrhea attend to out clinic labs of Assiut University hospital or admitted in gastroenterology, nephrology and oncology department of hospital during the study period.

Exclusion Criteria:

1. viral and bacterial causes of diarrhea
2. Patients who were already diagnosed as intestinal inflammatory disease as irritable bowel syndrome.
3. Autoimmune conditions, such as ulcerative colitis, Crohn's disease and coeliac disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: -Children presented with secretory diarrhea(acute watery diarrhea) attend to out clinic lab of Assiut University pediatric hospital or admitted in pediatric hospital(gastroenterology department) during the study period.
  2-adult patients having acute watery diarrhea attend to out clinic labs of Assiut University hospital or admitted in gastroenterology, nephrology and oncology department of hospital during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
percentage of patients with positive stool analysis for cryptosporidium | 2 days
  Use of microscopic examination and real time polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa M Abd elaziz, MD, Principal Investigator — Assuit University, Faculty of medicine
Locations (1):
- Heba gamal rashed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pawlowski SW, Warren CA, Guerrant R. Diagnosis and treatment of acute or persistent diarrhea. Gastroenterology. 2009 May;136(6):1874-86. doi: 10.1053/j.gastro.2009.02.072. Epub 2009 May 7. PMID 19457416